CLINICAL TRIAL: NCT06286163
Title: Neuroinflammatory Interactions of ATP and P2X3 Receptor in the Airways of Chronic Cough Patients: an Exploratory Study
Brief Title: Neuroinflammatory Interactions of ATP and P2X3 Receptor in the Airways of Chronic Cough Patients
Status: Recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: PA4099
Record Dates: First submitted 2024-02-22; First posted 2024-02-29 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Chronic Cough
MeSH Terms: conditions — Chronic Cough

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic Cough: History of chronic cough of at least 8 weeks' duration and should have been followed in the Cough Clinic for at least 6 months.
  Undergone a protocol with a diagnostic pathway as recommended by the ERS guidelines for management of cough.
  Would have either an identifiable cause for their cough that have failed therapies targeted towards the identified cause or classed as having chronic idiopathic cough where no identifiable cause has been found.
- Healthy: Healthy individuals, free of significant disease No history of asthma/rhinitis, No therapies, Baseline FEV1 ≥80% predicted with FEV1/FVC ratio >70% Non-smoker for at least the past 12 months with a pack history of ≤5 pack-years

SUMMARY:
This study is being done in order to understand what causes people to have a chronic cough, which is defined as a cough lasting for more than 8 weeks. The research team wish to find out whether there is any inflammation in the lungs of patients with chronic cough. The research team will also determine whether a suspected chemical produced in the body, called adenosine triphosphate (ATP) can be responsible for causing the chronic cough. In order to be able to find out what is abnormal in those who have a chronic cough, The research team will need to compare their results with those that do not have a chronic cough.

In this study, the research team will examine 10 participants who suffer from chronic cough and 8 individuals who do not have a chronic cough and are healthy.

DETAILED DESCRIPTION:
Background to problem Chronic cough is a very common clinical problem that is experienced by a large number of people and is a condition that can last for many years. It remains a difficult problem to treat by doctors because there is at present very poor understanding of what causes this condition of chronic cough. Consequently, the research team do not have much efficacious treatments for this common condition. Often, a cause for the cough can be identified by the doctor and treatment of the cause can help reduce or remove the cough. But in many instances, the cough may not be helped. In many cases also, the cause of the cough is not identified. These types of cough can be referred as being 'refractory' or 'idiopathic' or 'unexplained'.

Recently, the notion that chronic cough results from a state of hypersensitivity has been put forward to explain this condition. This has been put forward because those suffering from chronic cough often report that changes in ambient temperature, laughing, talking on the phone for more than a few minutes, aerosol sprays, or smoky atmospheres characteristically trigger bouts of coughing, indicating this state of hypersensitivity as a key common characteristic in this condition. Furthermore, this state of Cough Hypersensitivity Syndrome (CHS) could be caused by damage to the nerves (in the lungs and in the brain) by factors including viral infection, chemicals and inflammation. The nervous system controlling the sensitivity of the cough is necessarily complex and likely involves various molecules such as receptors and proteins that increase the sensitivity to cough.

Recently, a blocker of a receptor of a substance called Adenosine triphosphate (ATP), receptor P2X3, called AF-219 of Gefapixant has been shown to be extremely effective in suppressing the chronic cough of patients with an idiopathic cough, with a reduction in the number of coughs by 75% when compared to inactive drug 11. This is a very significant result because this study would suggest that this ATP receptor, P2X3, may play an important part in cough hypersensitivity syndrome. ATP is produced by cells and is the source of energy for cells needed for cellular functions such as movement of the cell and division of the cell.

Indeed, the academic community knows very little about the role of ATP and its receptor, P2X3, in chronic cough. First, it is possible that ATP may be released in greater amounts in chronic cough from activated or stressed cells in the airways, including nerves. ATP can cause inflammation and can be involved in the movement of inflammatory cells, production of oxygen free radicals by neutrophils and production of cytokines by inflammatory cells. ATP may induce a neuroimmune inflammatory response that could sensitise the peripheral nerves to cause this hypersensitivity. Through the PX3R, ATP can cause long-lasting allodynia through sensitisation of these receptors. Patients with chronic cough cough more to inhaled ATP compared to healthy subjectsparticipants.

Therefore, The research team want to show that:

1. ATP is released by cough stimuli and stimulates P2X3 receptors in the upper and lower airways
2. The increased sensory state of the peripheral sensory nerves leads to activation of P2X3 4 Together, these form the basis of cough hypersensitivity syndrome

ELIGIBILITY:
Inclusion Criteria:

- 1. For Normal non-smoking subject: Healthy individuals, free of significant disease No history of asthma/rhinitis, No therapies, Baseline FEV1 ≥80% predicted with FEV1/FVC ratio >70% Non-smoker for at least the past 12 months with a pack history of ≤5 pack-years

2. For chronic cough participants: History of chronic cough of at least 8 weeks' duration and should have been followed in the Cough Clinic for at least 6 months.

Undergone a protocol with a diagnostic pathway as recommended by the ERS guidelines for management of cough.

Would have either an identifiable cause for their cough that have failed therapies targeted towards the identified cause or classed as having chronic idiopathic cough where no identifiable cause has been found.

3. General Inclusion Criteria: Give written informed consent prior to participation in the study including all of its procedures. Comply with the requirements and restrictions listed in the consent form.

Male or female subject aged between 30 and 70 years old at screening. Able to complete the study and all measurements. Able to read, comprehend, and write at a sufficient level to complete study related materials.

Exclusion Criteria:

-

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who suffer from chronic cough and healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 18 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Presence of ATP in airways of idiopathic chronic cough patients and the localisation of P2X2/3 receptors in the airways | 18 months
  Measure ATP concentrations in exhaled breath condensate and use immunohistochemistry to identify P2X2/3 receptors in lung endobronchial biopsies.
Cough sensitivity and laryngeal sensitivity to exogenous ATP | 18 months
  Count the number of cough in response to capsaicin pre and post ATP exposure
Examine the effects of exogenous ATP on the inflammatory response in the upper and lower airways. | 18 months
  Count the number of immune cells in sputum and BALF pre and post ATP by microscopy

CONTACTS AND LOCATIONS:
Overall Officials: Kian Fan Chung, MD, Principal Investigator — Imperial College London
Locations (2):
- United Kingdom (2):
  - Royal Brompton & Harefield NHS Trust,, London
  - Royal Brompton Hospital, London

IPD SHARING:
Plan to Share IPD: No